CLINICAL TRIAL: NCT01629745
Title: Feasibility of Minimal Residual Disease (MRD) Determination in Pediatric B-Lineage ALL Using Deep Sequencing of the Immunoglobulin Heavy Chain Locus
Brief Title: Genetic Test in Detecting Minimal Residual Disease in Samples From Younger Patients Registered on the COG-AALL08B1 Trial
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B6; COG-AALL12B6 (Other: Children's Oncology Group); NCI-2012-01981 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: B-cell childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Testing for minimal residual disease in blood samples from patients with acute lymphoblastic leukemia may help doctors plan better treatment.

PURPOSE: This research trial studies a genetic test in detecting minimal residual disease in samples from younger patients registered on COG-AALL08B1 trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the feasibility of minimal residual disease (MRD) determination in pediatric B-lineage acute lymphoblastic leukemia (ALL) using deep sequencing of the immunoglobulin heavy chain locus.

OUTLINE: Archived blood and tumor tissue samples are analyzed for MDR using deep sequencing of immunoglobulin heavy chain locus. MDR quantification results are then compared with the flow cytometry reference methods used in COG studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples from patients registered on the Children Oncology Group (COG)-AALL08B1 protocol and stored in the Hematopathology Laboratory at the University of Washington

  * Pretreatment and after induction therapy samples

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Samples from patients registered on the Children Oncology Group (COG - AALL08B1)
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of deep sequencing of the immunoglobulin heavy chain locus in determining MRD in B-lineage ALL

CONTACTS AND LOCATIONS:
Overall Officials: Brent Wood, MD, PhD, Principal Investigator — Seattle Cancer Care Alliance